CLINICAL TRIAL: NCT06244043
Title: Human and Digital Support Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Thrive Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-1379; A171600 (Other: UW Madison); EDUC/COUNSELING PSYCH (Other: UW Madison)
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Depression; Anxiety
Keywords: meditation; app; HMP; Healthy Minds Program
MeSH Terms: conditions — Depression; Anxiety Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be informed which version of the introductory coaching session they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Initial Interventional Coaching Call Plus Email Support (Active Comparator)
  Interventions: Other: Initial Coaching Call; Other: Email Support; Other: Text Messages
- Initial Interventional Coaching Call No Email Support (Active Comparator)
  Interventions: Other: Initial Coaching Call; Other: Text Messages
- Initial Informational Coaching Call Plus Email Support (Active Comparator)
  Interventions: Other: Email Support; Other: Text Messages
- Initial Informational Coaching Call No Email Support (Active Comparator)
  Interventions: Other: Text Messages

INTERVENTIONS:
Other: Initial Coaching Call — Participant will receive initial coaching call with a team member. This coaching call will either be interventional (i.e., include content intended to prompt their adherence and benefit from the HMP app) or informational (i.e., include content intended to control for the time and attention of attending a coaching session, but not intended to provide specific benefits).
  Arms: Initial Interventional Coaching Call No Email Support; Initial Interventional Coaching Call Plus Email Support
Other: Email Support — Email-based support throughout study period
  Arms: Initial Informational Coaching Call Plus Email Support; Initial Interventional Coaching Call Plus Email Support
Other: Text Messages — All participants with receive text messages encouraging them to engage in the practices taught in the app.

SUMMARY:
The overall purpose of this study is to help determine how best to incorporate small amounts of human and digital support into a meditation app. 32 participants will be enrolled and can expect to be on study for up to 4 weeks.

DETAILED DESCRIPTION:
The overall purpose of this study is to help determine the feasibility and acceptability of incorporating small amounts of human and digital support into a meditation app. Ultimately, the investigators hope this work will help to develop digital tools that can reduce symptoms of depression and/or anxiety. The meditation app of interest is the Healthy Minds Program (HMP). The HMP app provides training in four pillars of well-being (Awareness, Connection, Insight, Purpose) through a combination of podcast-style didactic material and guided meditation practices.

Participants will be randomly assigned to receive or not receive an initial coaching call with a team member. Participants will also be randomly assigned to receive or not receive access to email-based support. All participants with receive text messages encouraging them to engage in the practices taught in the app.

Participants will complete a set of questionnaires at baseline and post-test (following the 4-week intervention period). Questionnaires and items will be selected from the set of questionnaires included in this application. The average length of time to complete questionnaires will be within 15 to 30 minutes. Participants will also receive short daily surveys.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18) who have recently downloaded the HMP app
* Elevated symptoms of depression and/or anxiety

  * Patient Health Questionnaire - 9 (PHQ-9) ≥ 5
  * General Anxiety Disorder - 7 (GAD-7) ≥ 5

Exclusion Criteria:

* Current suicidal or self-harm ideation (PHQ-9 item 9 > 0)
* Current or past psychotic disorder
* Current of past bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Study completion rate | Baseline to 4 weeks (post-intervention)
  Percentage of participants completing pre- and post-test measures
Daily diary completion rate | Baseline to 4 weeks (post-intervention)
  Percentage of daily assessments completed
Acceptability of Intervention Score | 4 weeks (post-intervention)
  12-item survey scored from 1 - 5 where higher scores indicate more acceptability.
Modified System Usability Scale Score | 4 weeks (post-intervention)
  10-item survey scored from 1-5 where higher scores indicate more usability.

OTHER OUTCOMES:
Attitudes Towards Psychological Online Interventions Score | 4 weeks (post-intervention)
  16-item survey scored from 1 - 5 where higher scores indicate more positive attitude in each of 4 domains: skepticism, confidence, threat, anonymity.
Determinants of Meditation Practice Inventory Score | baseline (pre-intervention)
  12-item survey scored from 1 - 5 where lower scores indicate lower perceived barriers to meditation practice in each of 4 domains; benefit, knowledge, pragmatic, cultural.
Patient Health Questionnaire - 9 (PHQ-9) Score | baseline (pre-intervention), 4 weeks (post-intervention)
  9-item survey scored from 0-27 where higher scores indicate increased depression.
PROMIS Meaning and Purpose Score | baseline (pre-intervention), 4 weeks (post-intervention)
  Computer adaptive survey scored from 1-5 where higher scores indicate higher sense of meaning and purpose.
Digital Working Alliance Inventory (D-WAI) Score | 4 weeks (post-intervention)
  6-item survey scored from 1-7 where higher scores indicate increased trust in the app in each of three domains: goals, tasks, bond.
Five Facet Mindfulness Questionnaire (FFMQ): Awareness Score | baseline (pre-intervention), 4 weeks (post-intervention)
  8-item survey scored from 1-5 where higher scores indicate lower levels of awareness.
General Anxiety Disorder -7 (GAD-7) Score | screening, 4 weeks (post-intervention)
  7-item survey scored from 0-21 where higher scores indicate increased anxiety.
Mindfulness Adherence Questionnaire: Minutes of meditation per week | 4 weeks (post-intervention)
  Minutes of meditation practice completed per week
Mindfulness Adherence Questionnaire Score | 4 weeks (post-intervention)
  10-item survey scored from 0-6 where higher scores indicate higher quality meditation practice in two domains: formal practice, informal practice.
Healthy Minds Index Score | baseline (pre-intervention), 4 weeks (post-intervention)
  17-item survey scored from 0-4 where higher scores indicate healthier attitude in each of 4 domains: awareness, connection, insight, purpose.
NIH Toolbox: Loneliness Score | baseline (pre-intervention), 4 weeks (post-intervention)
  5-item survey scored from 1-5 where higher scores indicate increased loneliness.
Growth Mindset Scale for Well-Being Score | baseline (pre-intervention), 4 weeks (post-intervention)
  3-item survey scored from 1-6 where higher score lower growth mindset.
Experiences Questionnaire Decentering Score | baseline (pre-intervention), 4 weeks (post-intervention)
  11-item survey scored from 1-5 where higher scores indicate higher levels of decentering.
Daily Diary Assessment Question Scores | daily from baseline to post-test (week 4)
  9-items administered in the morning scored from 1 (not at all) to 5 (very much) for domain: mindfulness, decentering, connection, purpose, depression, anxiety, stress, rumination, motivation.
  11-items administered in the evening scored from 1 (not at all) to 5 (very much) for domain: mindfulness, decentering, connection, purpose, depression, anxiety, happy event, stressor exposure item, rumination, informal practice item, formal practice item.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No